CLINICAL TRIAL: NCT01166529
Title: Endoscopic Ultrasound (EUS)-Guided Celiac Plexus Neurolysis (CPN) in the Management of Pain in Abdominal Non-pancreatic Malignancies
Brief Title: Endoscopic Ultrasound-guided Celiac Plexus Neurolysis in the Management of Pain in Abdominal Non-pancreatic Malignancies
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to identify appropriate patients.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Rajesh Keswani, Asssociate Professor, Northwestern University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NU protocol #0917 (eIRB 20311)
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Pain; Cancer
MeSH Terms: conditions — Pain; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EUS-CPN (Experimental)
  Interventions: Procedure: EUS-guided Celiac Plexus Neurolysis

INTERVENTIONS:
Procedure: EUS-guided Celiac Plexus Neurolysis — All patients will receive anesthesia. The linear echo-endoscope will be advanced into the proximal stomach. It will be noted whether the tumor is seen in the celiac axis, if there is flow in the celiac artery, and if the celiac ganglia are seen. The celiac ganglia will be injected directly with 10cc of 0.25% bupivicaine followed by 10cc of 98% dehydrated alcohol. If the celiac ganglia cannot be identified, the posterior and anterior aspects of celiac artery take-off will be injected in a similar manner (twice the volume). Flow in the celiac axis will be confirmed. All injections will be performed with a standard EUS injection needle made especially for CPN . Prior to injection, aspiration will be performed through the needle to ensure that no blood is aspirated.

SUMMARY:
Celiac plexus neurolysis (CPN) has been performed for nearly 100 years to alleviate the abdominal pain associated with pancreatic malignancy and other conditions, and is usually undertaken at a late stage in the disease process, when analgesic options have been largely exhausted or have led to significant and often unacceptable side effects. Until recently, CPN was most commonly performed under radiographic guidance; however, in the last 10 years, CPN has been routinely performed under endoscopic ultrasound (EUS) guidance. Several case series have demonstrated the efficacy and safety of this technique when used to treat the pain associated with pancreatic malignancy and/or chronic pancreatitis. However, the efficacy of EUS-guided CPN in the treatment of pain related to non-pancreatic malignancies has yet to be described. The goal of this study is to assess the efficacy of EUS-guided CPN in the management of pain in patients with abdominal non-pancreatic malignancies. Our hypothesis is that EUS-guided CPN will provide adequate pain relief in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an unresectable, non-pancreatic malignancy, including gastric, small intestinal, or proximal colonic malignancies, as well as malignancies of the liver and bile ducts (based on above celiac plexus innervations)
* Pain directly related to the primary malignant process, as determined by the referring oncologist
* Pain determined to be refractory to standard medical therapy, or when the medical therapy is ineffective due to certain limitations (such as severe constipation), as determined by the referring oncologist
* Willingness to undergo EUS-guided CPN
* Age > 18 years
* ECOG performance status of grades 0-3 [7]
* The patient will need to sign informed consent prior to inclusion in this study

Exclusion Criteria:

* Unable or unwilling to undergo an EUS-guided CPN
* Contraindication to anesthesia, as determine during the preoperative clearance process
* Refractory coagulopathy (INR > 1.5) or thrombocytopenia (platelet count < 50,000), or aspirin and/or clopidogrel use within 7 days of procedure
* Current pregnancy
* Prior celiac plexus block/neurolysis
* Allergy to local anesthetics
* ECOG performance status of grade 4 or higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Difference between the mean pain score prior to and 1 month after the procedure, as determined by the Brief Pain Inventory (BPI) | 1 month
  The BPI will be filled out just prior to and 1 month after the procedure to assess the difference in the mean pain score after the procedure

SECONDARY OUTCOMES:
Difference in mean pain scores before and at 1 day after the procedure, 7 days after the procedure, 14 days after the procedure, and at 2 months after the procedure, as determined by the Brief Pain Inventory (BPI). | 2 months
  The BPI will be filled out just prior to the procedure and after the procedure at the above intervals (up to 2 months) to assess the difference in the mean pain scores after the procedure.
Difference in the mean 'level of interference of pain with daily life' score, as determined by the Brief Pain Inventory (BPI). This score will be determined before and after the procedure, determined at the same intervals as mean pain scores. | 2 months
Narcotic use over a 24-hour period will be documented each time the Brief Pain Inventory (BPI) is completed | 2 months
  Names, doses, and quantity of pain medications will be reported and converted to an equianalgesic dose (mg/day) of orally administered morphine. The difference in equianalgesic doses (mg/day) will be determined at the same intervals as mean pain scores.

CONTACTS AND LOCATIONS:
Overall Officials: Raj N Keswani, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Christo PJ, Mazloomdoost D. Interventional pain treatments for cancer pain. Ann N Y Acad Sci. 2008 Sep;1138:299-328. doi: 10.1196/annals.1414.034. PMID 18837908
- [Background] Chak A. What is the evidence for EUS-guided celiac plexus block/neurolysis? Gastrointest Endosc. 2009 Feb;69(2 Suppl):S172-3. doi: 10.1016/j.gie.2008.12.022. No abstract available. PMID 19179150
- [Background] Penman ID, Rosch T; EUS 2008 Working Group. EUS 2008 Working Group document: evaluation of EUS-guided celiac plexus neurolysis/block (with video). Gastrointest Endosc. 2009 Feb;69(2 Suppl):S28-31. doi: 10.1016/j.gie.2008.11.004. No abstract available. PMID 19179165
- [Background] Puli SR, Reddy JB, Bechtold ML, Antillon MR, Brugge WR. EUS-guided celiac plexus neurolysis for pain due to chronic pancreatitis or pancreatic cancer pain: a meta-analysis and systematic review. Dig Dis Sci. 2009 Nov;54(11):2330-7. doi: 10.1007/s10620-008-0651-x. Epub 2009 Jan 10. PMID 19137428
- [Background] Daut RL, Cleeland CS, Flanery RC. Development of the Wisconsin Brief Pain Questionnaire to assess pain in cancer and other diseases. Pain. 1983 Oct;17(2):197-210. doi: 10.1016/0304-3959(83)90143-4. PMID 6646795
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009